CLINICAL TRIAL: NCT00366184
Title: Influencing Motor Performance in Patients With Stroke by Combined Theta Burst Stimulation and Carbidopa-Levodopa
Brief Title: Influence of Theta Burst Stimulation and Carbidopa-Levodopa on Motor Performance in Stroke Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060225; 06-N-0225
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-05-26

CONDITIONS: Stroke
Keywords: Neuromodulation; Stroke; Motor Cortex; Motor Learning; L-Dopa; Transcranial Magnetic Stimulation; Levodopa; Healthy Volunteer; HV
MeSH Terms: conditions — Stroke

SUMMARY:
This study will examine whether transcranial magnetic stimulation (TMS) of the brain used in combination with carbidopa-levodopa is more effective in temporarily improving the speed of hand movement in stoke patients than TMS alone. In TMS, a wire coil is held on the patient's scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. The effect of TMS on the muscles is detected with small metal disk electrodes taped to the skin of the arms or legs. Carbidopa-levodopa is a medication usually used to treat Parkinson's disease, but it may improve the effect of theta burst stimulation.

Two kinds of TMS are used in this study. In single-pulse TMS one or two pulses are delivered at a time in order to measure brain activity at that moment. In repetitive TMS (rTMS), a series of pulses are given in short bursts, temporarily altering brain activity. The type of rTMS used in this study is called theta burst stimulation.

Healthy normal volunteers and people who had a stroke 6 months or more before entering the study may be eligible to participate. All candidates must be between 18 and 90 years of age. Stroke patients must have had significant hand weakness and made a moderate or good recovery and must be able to move either the thumb or the wrist on the affected hand reasonably well. Normal volunteers must be right-handed.

Participants complete the testing for this study in four main sessions scheduled at least a week apart and five short follow-up sessions. At each main session, participants take either a carbidopa-levodopa tablet or a placebo (a look-alike inactive substance). Stroke patients have their arm and hand function assessed using two tests. One requires them to insert pegs into holes; the other includes writing, lifting various objects, and performing activities like turning pages, feeding or stacking checkers.

All subjects complete a questionnaire regarding their mood and alertness and then perform tests of thumb or wrist movement. For this test, a small electrical stimulus is applied to the side of the hand and the subject must respond to the stimulus as quickly as possible by making a thumb or wrist movement. This is repeated several times over about 3 minutes. A second test follows in which the subject moves the thumb or wrist in response to a beep from a speaker. This test is repeated several times over about 8 minutes. Some measurements are taken using single-pulse TMS during the beginning, middle and end of this test. In two of the four sessions, theta burst stimulation is applied after the single-pulse TMS and in the other two sessions, sham theta burst stimulation is applied.

Five follow-up sessions are scheduled one day after each main session and one week following the final one. In these sessions, subjects perform an abbreviated form of the thumb movement tests.

DETAILED DESCRIPTION:
OBJECTIVE:

Theta Burst Stimulation (TBS) is a type of sub-threshold repetitive Transcranial Magnetic Stimulation (rTMS) which has effects on the excitability of human motor cortex that outlast stimulation by up to an hour. TBS also affects performance of a motor task for up to 30 minutes after stimulation in healthy subjects, and improves reaction times (and increases corticospinal excitability) in patients with chronic stroke (Talelli 2005). The advantages of TBS over other non-invasive brain stimulation strategies are its low intensity, short duration of application and long lasting effects.

The spectrum of behavioral effects investigated is so far modest. Evidence is accumulating that dopaminergic agents enhance synaptic plasticity (Otani 1998) and improve motor training in healthy humans (Meintzchel 2005). After stroke, Carbidopa-Levodopa has also enhanced the response to physiotherapy and motor learning (Scheidtmann 2001, Floel 2005). This protocol aims to test the hypothesis that Carbidopa-Levodopa may enhance the beneficial effect of TBS on reaction times in patients with chronic stroke.

STUDY POPULATION:

We plan to investigate 18 patients with motor impairment more than 6 months after ischemic stroke, and 10 healthy volunteers. Approval is sought for a total of 28 patients and 30 healthy volunteers to account for possible dropouts and pilot experiments (described below).

DESIGN:

Each subject will be asked to participate in 4 sessions, at least a week apart. The experiment will test simple reaction times in the thumb or wrist of the paretic hand before and 7 minutes after either genuine or sham TBS. This will be followed by a measure of motor learning, using a well-characterized paradigm (Muellbacher 2001), which involves optimizing an externally paced ballistic thumb (or wrist) movement, and TMS measurement of corticospinal excitability. Performance of the learned task will be further assessed (and TMS measures made) at 2 hours, 1 day and 1 week following the training session. The experimental design for the four sessions will be 2x2 with TBS/sham and Carbidopa-Levodopa/placebo. For TBS, the patient will be given 3 minutes of either genuine or sham TBS to the hand representation of the motor cortex (Huang 2005). For Carbidopa-Levodopa/placebo, identical preparations from the NIH pharmacy will be given 1 hour beforehand. TBS has previously been used in 72 healthy subjects (7 studies) in Europe and in 10 patients with chronic stroke (2 studies) in the Lead Associate Investigator's lab in London. No side effects or seizures have been reported. Ten normal volunteers will be studied first to optimize experimental settings.

OUTCOME MEASURES:

The primary outcome measure will be reaction times. Improvement in peak acceleration in the learning task will constitute a secondary measure. We expect to see improved reaction times with genuine TBS (vs. sham) and will look for an interaction whereby Carbidopa-Levodopa may enhance this effect (vs. placebo). This would suggest that synergy between dopaminergic modulation and TBS may show promise to produce clinical gains after stroke.

ELIGIBILITY:
* INCLUSION CRITERIA:

PATIENTS:

* Age 18 - 90
* Ischemic cerebral infarction more than 6 months prior to testing not involving cortical motor areas
* Initial severe paresis (MRC Grade 2 or less in hand muscles) with considerable motor recovery
* Ability to make ballistic thumb abduction or wrist extension movements in the affected hand

HEALTHY SUBJECTS:

* Age 18 - 90
* Right handed
* Able to concentrate and to perform the tasks required

EXCLUSION CRITERIA:

PATIENTS:

* More than one ischemic stroke, or any hemorrhagic stroke
* Large cortical stroke
* Significant cognitive impairment, defined as a Mini Mental State Examination score of 23 or less
* History of seizures or other neurological illness (except stroke)
* History of alcohol or drug abuse
* Inability to make necessary thumb abduction or wrist extension movements
* Current or recent use of neuroleptic medication, tricyclic anti-depressants or monoamine oxidase inhibitors
* History of narrow angle glaucoma
* Contraindications to TMS - presence of cardiac pacemaker, intracardiac lines, implanted pumps or stimulators, or metal objects inside the eye or skull
* Pregnancy (as the effects of TBS on the fetus are as yet unknown)
* Uncontrolled medical (e.g. cardiovascular disease expressed as uncontrolled arrhythmias, shortness of breath, or overt signs of severe peripheral edema at the initial neurological exam, severe rheumatoid arthritis, arthritic joint deformity, active cancer or renal disease), or psychiatric problems (defined as having received medical treatment from a psychiatrist).

HEALTHY SUBJECTS:

* Contraindications to TMS (as above)
* Pregnancy (see above)
* History of seizures or other neurological illness
* History of alcohol or drug abuse
* History of depression / psychiatric illness requiring use of anti-psychotic drugs or anti-depressants
* Current or recent use of neuroleptic medication, tricyclic anti-depressants or monoamine oxidase inhibitors
* History of narrow angle glaucoma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-08-08; Study Completion 2010-05-26

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Conforto AB, Kaelin-Lang A, Cohen LG. Increase in hand muscle strength of stroke patients after somatosensory stimulation. Ann Neurol. 2002 Jan;51(1):122-5. doi: 10.1002/ana.10070. PMID 11782992
- [Background] Di Lazzaro V, Pilato F, Saturno E, Oliviero A, Dileone M, Mazzone P, Insola A, Tonali PA, Ranieri F, Huang YZ, Rothwell JC. Theta-burst repetitive transcranial magnetic stimulation suppresses specific excitatory circuits in the human motor cortex. J Physiol. 2005 Jun 15;565(Pt 3):945-50. doi: 10.1113/jphysiol.2005.087288. Epub 2005 Apr 21. PMID 15845575
- [Background] Donoghue JP. Plasticity of adult sensorimotor representations. Curr Opin Neurobiol. 1995 Dec;5(6):749-54. doi: 10.1016/0959-4388(95)80102-2. PMID 8805413